CLINICAL TRIAL: NCT06893939
Title: Limited Versus Extended Trophic Feeding (LET-FEED) Trial
Acronym: LET-FEED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Alabama at Birmingham (Other); Baylor College of Medicine (Other); University of South Florida (Other); University of Oklahoma (Other); St. Joseph's Medical Center (Unknown)
Responsible Party: Principal Investigator, Gregory C. Valentine, MD MED FAAP, Associate Professor, Department of Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00021132
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Length of Stay; Mortality
Keywords: Feeding; Nutrition; Prematurity; Very preterm; Trophic; Trophic feeds; Trophic feeding; enteral feeds; sepsis
MeSH Terms: conditions — Sepsis; Premature Birth

STUDY DESIGN:
Masking Description: This will be an open label trial as it relates to do different feeding approaches preventing masking/blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended Trophic Feeding (Active Comparator): Advancing enteral feeds after 3 days of trophic feeds of 20-25 mL/kg birthweight/day. Advancement of enteral feeds will be by approximately 30 mL/kg birthweight/day after 3 days of trophic feeds. Advancement will occur until achieving at least 140 mL/kg birthweight/day of enteral feeds. Enteral feeds will consist of parent's own milk or donor human milk.
  Interventions: Other: Extended Trophic Feeds (3 days of trophics)
- Limited Trophic Feeds (Experimental): Advancing enteral feeds after 1 day of trophic feeds of 20-25 mL/kg birthweight/day. Advancement of enteral feeds will be by approximately 30 mL/kg birthweight/day until achieving at least 140 mL/kg birthweight/day of enteral feeds. Enteral feeds will consist of parent's own milk or donor human milk.
  Interventions: Other: Limited Trophic Feeds (1 day of trophic feeds)

INTERVENTIONS:
Other: Limited Trophic Feeds (1 day of trophic feeds) — Advancing enteral feeds after 1 day of trophic feeds of 20-25 mL/kg birthweight/day. Advancement of enteral feeds will be by approximately 30 mL/kg birthweight/day until achieving at least 140 mL/kg birthweight/day of enteral feeds. Enteral feeds will consist of parent's own milk or donor human milk.
  Other Names: Limited Trophic Feeds
  Arms: Limited Trophic Feeds
Other: Extended Trophic Feeds (3 days of trophics) — Advancing enteral feeds after 3 days of trophic feeds of 20-25 mL/kg birthweight/day. Advancement of enteral feeds will be by approximately 30 mL/kg birthweight/day after 3 days of trophic feeds. Advancement will occur until achieving at least 140 mL/kg birthweight/day of enteral feeds. Enteral feeds will consist of parent's own milk or donor human milk.
  Arms: Extended Trophic Feeding

SUMMARY:
Study Hypothesis/Question In infants born very preterm, advancing enteral feeds after 24 hours from birth (limited trophic feeds) versus after 72 hours (extended trophic feeds) reduces the risk of all-cause late onset sepsis (LOS) without increasing the risk of other adverse outcomes.

Study Design Type This is a multi-center, open-label, parallel-group, individual randomized controlled trial comparing two different trophic feeding regimens in preterm infants born between 25w0d and 31w6d. These infants will be randomly assigned to either the intervention group, receiving limited trophic feeding (20 to 25 mL/kg/day for one day) or the control group, receiving extended trophic feeding (20 to 25 mL/kg/day for three days) prior to advancing enteral feeds until full feeding volume (140 mL/kg/day) is achieved.

Eligibility Criteria Preterm infants with gestational ages between 25 0/7 and 31 6/7 weeks and a birthweight of <1500 grams who are admitted to six participating neonatal units will be eligible for inclusion. Infants with <5th percentile for weight at birth, vasopressor use within first 24 hours of life major congenital/genetic anomalies affecting enteral feeding, growth, or mortality, and those with a terminal illness in which decisions to withhold or limit support have been made will be excluded. Infants of parents or legal guardians who are unable to provide consent within 36 hours of birth will also be excluded.

Study Intervention/Methods Written parental informed consent will be obtained prenatally or within the first 36 hours of birth. Infants will be randomized to receive limited trophic feeds of 24 to 36 hours or extended trophic feeds for 72 hours prior to the advancement of enteral feeds. Infants will be fed parent's own milk (POM) with donor human milk as the alternative if POM is unavailable.

Primary Outcome Late-onset sepsis, defined as positive blood, urine, and/or cerebrospinal fluid (CSF) cultures in the presence of compatible clinical signs of sepsis, occurring after postnatal day 3 and before hospital discharge, and treated with antibiotics for 5 days or more.

Secondary Outcome(s) The trial will assess various secondary outcomes including length of hospital stay, all-cause in-hospital mortality, duration of IV fluids and central line utilization, necrotizing enterocolitis (Bell's stage IIa or higher), severe intraventricular hemorrhage (grade III or IV either unilaterally or bilaterally), bronchopulmonary dysplasia (oxygen requirement or positive pressure ventilation at 36 weeks corrected gestational age), or retinopathy of prematurity requiring intervention. Additionally, growth metrics throughout hospitalization will be evaluated using change in weight, length, and head circumference z-scores from birth to 36 weeks' corrected gestational age between infants in the limited and extended trophic feeding groups.

DETAILED DESCRIPTION:
Up to 30% of all very preterm (VP; defined as those born before 32 weeks' gestation) newborns born within the United States develop late onset sepsis (LOS), a life-threatening infection that occurs after 72 hours from birth. LOS is the leading cause of morbidity in all very preterm newborns. VP newborns who develop LOS have significantly lower survival rates (adjusted risk ratio [aRR] 0.89, 95% confidence interval [CI] 0.87-0.90), 32% increased risk of being discharged on oxygen (aRR 1.32, 95% CI 1.26-1.38), 288% increased risk of needing a tracheostomy (aRR 2.88, 95% CI 2.47-3.37), and a 209% increased risk of requiring a gastrostomy tube (aRR 2.09, 95% CI 1.93-2.57).27 Thus, clinical practices that can reduce LOS are critically important to ensure VP newborns not only survive, but thrive, living lives free of disability or impairment.

One of the most protective factors in preventing LOS is an exclusive human milk-based diet. Common clinical practice for VP newborns includes starting human milk-based enteral feeds at approximately 20 mL/kg/day (e.g. "trophic feeds") and then progressively advancing the volume of enteral feeds daily until reaching a sufficient quantity to achieve adequate hydration and nutrition (e.g. "full feeds"). While enteral feeds are being advanced, VP newborns receive additional supplementary fluids and nutrition via intravenous (IV) infusions. Yet, any indwelling catheter to provide IV nutrition inherently increases the risk of LOS because the catheter breaches the newborn's protective skin barrier, thereby increasing risk of invasive infection from skin microbes.

One way to reduce the need for IV fluids is to initiate enteral human milk feeds earlier and advance feeds faster, thereby limiting the duration of indwelling IV catheters. An additional benefit of this approach is that early introduction of human milk prevents dysbiosis of the neonatal microbiome that is associated with LOS. By preventing the growth of harmful, pathogenic, sepsis-causing bacteria within the gut of VP newborns, these newborns have overall less risk of developing LOS. Yet, these benefits are with an exclusive human milk-based diet as meta-analyses and systematic reviews have demonstrated that feeding formula significantly increases the risk of necrotizing enterocolitis (NEC), a devastating inflammatory process within the gastrointestinal system that is associated with a 30-50% mortality rate.

A Gerber-funded (AA Salas PI, novice research award), pilot randomized trial that compared early versus delayed progressive feeding in 60 extremely preterm infants born at the University of Alabama Hospital showed that early progressive feeding reduced the need for central venous access (p=0.0001) and parenteral nutrition by 4 days (p=0.0005). Culture-proven sepsis (10% vs. 27%; p= 0.18) tended to be lower in the early progressive feeding group but did not reach statistical significance due to the limited power and sample size of the study.

Thus, the natural next question is whether early progression of enteral feeds in a multi-center trial improves clinical outcomes, namely prevention of invasive infection, without increased risk of adverse outcomes including mortality. The lack of multi-center clinical trials evaluating faster advancement of enteral feeds to full volume feeds has left clinicians with uncertainty about the risks and benefits of this approach and resulted in a lack of uniformity in clinical practice. This has led to significant differences in how VP newborns are fed across the US and globally, with some centers initiating and advancing feeds within the first few hours after birth and others continuing small volume "trophic" feeds without any advancement until day 4 after birth. Thus, clinicians caring for VP newborns are in dire need of evidence to determine the optimal feeding advancement strategy to improve their short- and long-term outcomes.

Study Population:

Investigators will enroll 350 very preterm infants born at 25 0/7 to 31 6/7 weeks' gestation admitted to the six participating neonatal intensive care units. All newborns will be eligible for this study without regards to gender, ethnicity, race, socioeconomic status, or language spoken. This study population has been selected based on the frequency of newborn admissions, sepsis, and overall mortality observed at these gestational ages. The participating centers include: (1) St. Joseph's Medical Center (Tacoma, WA), (2) Baylor College of Medicine (Houston, TX), (3) University of Alabama (Birmingham, AL), (4) University of South Florida (Tampa, FL), and (5) University of Oklahoma (Oklahoma City, OK).

Consent and Randomization:

To ensure timely enrollment, written informed consent will be obtained no later than 36 hours following birth, with a goal of enrollment within 24 hours of birth or prenatally. Identification of potential participants will prompt a visit from a study team member, who will meet with the parent(s) in their room or the baby's room to explain the study. During this meeting, the risks and benefits associated with participation will be thoroughly discussed, and ample time will be allocated for the parents to ask any questions they may have. The consent will include that the newborn will be fed parent's own milk as the prioritized enteral feed with donor milk as the alternative if POM is of insufficient quantity.

Importantly, participants will be assured that their infant will receive all necessary treatments irrespective of their involvement in the study. The process of randomization will then determine the assignment of each participant to their respective study group.

Participants will be randomly assigned to one of the study groups following computer generated random-block sequences. The University of Washington will develop the sequence and implement stratified randomization by gestational age using a computerized central telephone system. Twin and multiple infants will be randomized individually.

Study Intervention and Active Comparator:

After consenting, information about the pregnancy and participating infant will be collected, including contact information for the parent(s), race/ethnicity, medical history, family history, education level, employment status, marital status, and other information to assess baseline characteristics of study participants.

All consented and enrolled infants will be randomly assigned to receive either limited trophic feeds of 24 hours or extended trophic feeds of 72 hours after birth prior to the advancement of enteral feeds. Given that IV fluids and parenteral nutrition need to be ordered up to 12 hours prior to the implemented change, investigators have included a 12-hour period of advancement (24 to 36 hours versus 72 to 84 hours after birth) to account for these logistics and ensure the generalizability of the trial's findings. Feeding volumes will be advanced by 25 to 30 mL/kg/day until full feeds (140 mL/kg/day) are reached within two weeks of birth.

All participating centers will provide parent's own milk as the prioritized feed, with human donor milk provided inn cases where POM is not available in sufficient quantities. Preterm formula will not be used. The trial will recommend that fortification occurs once enteral feeding volumes of 40 to 60 mL/kg/day or higher are achieved and that IV catheters will be removed once the newborn is above 120 mL/kg/day of enteral feeds.

Deviations from the feeding protocol will be allowed if signs of feeding intolerance are present before establishment of full enteral feeding. Feeding intolerance will be defined as an interruption or cessation of enteral feeds for a period greater than 12 hours for abnormal abdominal examination within 14 days of birth. Information will also be collected on the percentage of enteral feeds that had a >50% reduction in planned volume over each 24-hour period to serve as an additional metric of feeding intolerance.

The primary outcome will be culture-proven late onset sepsis. Culture-proven LOS will be defined as positive blood, urine, and/or cerebrospinal fluid (CSF) cultures in the presence of compatible clinical signs of sepsis, occurring between postnatal day 3 and hospital discharge, necessitating treatment with antibiotics for 5 days or more.

ELIGIBILITY:
Inclusion Criteria:

* <1500 gram birthweight
* 25w0d-31w6d at birth
* Consent to feed donor milk when parent's own milk is not available or of insufficient quantity

Exclusion Criteria:

* <5th percentile for weight at birth (Fenton growth curve)
* Parent or legal guardian unable to provide consent within 36 hours after birth
* Congenital anomaly affecting decisions on enteral feedings (e.g. gastroschisis, omphalocele, congenital diaphragmatic hernia, congenital heart disease, etc.)
* Known genetic condition affecting growth, feeding, or mortality
* Vasopressor use within first 24 hours after birth (not including hydrocortisone)
* Considered terminally ill

Ages: 0 Hours to 36 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Late Onset Sepsis | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Defining LOS: For the purposes of this study, a positive finding of LOS will be defined as the following: a body fluid culture (e.g. blood, urine, CSF) that returns positive, obtained in the presence of compatible clinical signs of sepsis (e.g. hypotension, apnea/bradycardia, increasing oxygen requirements, increasing metabolic acidosis, lactic acidosis, hypoglycemia, hyperglycemia, etc.) occurring after 72 hours from birth and before hospital discharge that was treated with antibiotics for a minimum of 5 days.

SECONDARY OUTCOMES:
All-Cause In-Hospital Mortality | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  all-cause in-hospital mortality
Duration of parenteral nutrition | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Days of parenteral nutrition during hospitalization
Duration of Central Venous Access | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Days of central venous access throughout hospitalization
Length of hospitalization | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Length of hospitalization (days)
Time to reach full enteral feeding volumes | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Full enteral feeding volumes defined as ≥120 mL/kg birthweight/day
Number of culture-proven late onset sepsis episodes | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Will be assess per participant throughout hospitalization
Type of late-onset sepsis | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Hematogenous/sepsis, urinary tract infection, meningitis, combination, or other
Necrotizing Enterocolitis | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Modified Bell's stage IIa or higher
Spontaneous Intestinal Perforation (SIP) | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  SIP diagnosed during hospitalization
Severe Intraventricular Hemorrhage (IVH) | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Defined as Grade III or IV unilaterally or bilaterally
Bronchopulmonary Dysplasia | At 36 weeks corrected gestational age
  Defined as needing supplemental oxygen or non-invasive administration of positive pressure, or invasive ventilation at 36 weeks corrected gestational age
Retinopathy of Prematurity requiring Intervention | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Medical or surgical intervention
Patent Ductus Arteriosus Requiring Intervention | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Medical or surgical intervention (not including prophylactic)
Type of pathogen detected in culture-positive late-onset sepsis | Through study completion, the end of NICU hospitalization, an average of 40 weeks' gestation
  Bacteria, fungal, or viral pathogen detected in any culture-positive late-onset sepsis event detected after 72 hours from birth and during hospitalization
Change in Z-score of weight | From admission to 36 weeks corrected gestational age
  From birth to 36 weeks corrected gestational age weight Z-score change
Change in Z-score of length | From admission to 36 weeks corrected gestational age
  From birth to 36 weeks corrected gestational age length Z-score change
Change in Z-score of head circumference | From admission to 36 weeks corrected gestational age
  From birth to 36 weeks corrected gestational age head circumference Z-score change

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Valentine, Principal Investigator — University of Washington
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Florida, Tampa, Florida
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington
  - St. Joseph's Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers if a scientifically sound and reasonable plan is provided to the study team investigators and Co-PIs. A data sharing or transfer use agreement may be required per institutional policy if sharing of data occurs.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified data will be shared with researchers requesting access to the data if they have a scientifically sound and reasonable plan. The data will be shared within 6-12 months of receiving the request by the researchers and a determination is made.
Access Criteria: Deidentified data will be shared with researchers requesting access to the data if they have a scientifically sound and reasonable plan. The data will be shared within 6-12 months of receiving the request by the researchers and a determination is made. The data will be transferred via a HIPAA secure format.

REFERENCES:
- [Background] Salas AA, Li P, Parks K, Lal CV, Martin CR, Carlo WA. Early progressive feeding in extremely preterm infants: a randomized trial. Am J Clin Nutr. 2018 Mar 1;107(3):365-370. doi: 10.1093/ajcn/nqy012. PMID 29529231
- [Background] Higgins BV, Baer RJ, Steurer MA, Karvonen KL, Oltman SP, Jelliffe-Pawlowski LL, Rogers EE. Resuscitation, survival and morbidity of extremely preterm infants in California 2011-2019. J Perinatol. 2024 Feb;44(2):209-216. doi: 10.1038/s41372-023-01774-6. Epub 2023 Sep 9. PMID 37689808
- [Background] Perez KM, Strobel KM, Hendrixson DT, Brandon O, Hair AB, Workneh R, Abayneh M, Nangia S, Hoban R, Kolnik S, Rent S, Salas A, Ojha S, Valentine GC. Nutrition and the gut-brain axis in neonatal brain injury and development. Semin Perinatol. 2024 Aug;48(5):151927. doi: 10.1016/j.semperi.2024.151927. Epub 2024 Jun 13. PMID 38897828
- [Background] Ohlin A, Bjorkman Hjalmarsson L. In neonatal sepsis every catheter matters. Pediatr Res. 2021 Sep;90(3):506-507. doi: 10.1038/s41390-021-01533-3. Epub 2021 Apr 17. No abstract available. PMID 33866330
- [Background] Singer JR, Blosser EG, Zindl CL, Silberger DJ, Conlan S, Laufer VA, DiToro D, Deming C, Kumar R, Morrow CD, Segre JA, Gray MJ, Randolph DA, Weaver CT. Preventing dysbiosis of the neonatal mouse intestinal microbiome protects against late-onset sepsis. Nat Med. 2019 Nov;25(11):1772-1782. doi: 10.1038/s41591-019-0640-y. Epub 2019 Nov 7. PMID 31700190
- [Background] Stewart CJ, Embleton ND, Marrs ECL, Smith DP, Fofanova T, Nelson A, Skeath T, Perry JD, Petrosino JF, Berrington JE, Cummings SP. Longitudinal development of the gut microbiome and metabolome in preterm neonates with late onset sepsis and healthy controls. Microbiome. 2017 Jul 12;5(1):75. doi: 10.1186/s40168-017-0295-1. PMID 28701177
- [Background] Lee CC, Feng Y, Yeh YM, Lien R, Chen CL, Zhou YL, Chiu CH. Gut Dysbiosis, Bacterial Colonization and Translocation, and Neonatal Sepsis in Very-Low-Birth-Weight Preterm Infants. Front Microbiol. 2021 Oct 7;12:746111. doi: 10.3389/fmicb.2021.746111. eCollection 2021. PMID 34690993
- [Background] Quigley M, Embleton ND, Meader N, McGuire W. Donor human milk for preventing necrotising enterocolitis in very preterm or very low-birthweight infants. Cochrane Database Syst Rev. 2024 Sep 6;9(9):CD002971. doi: 10.1002/14651858.CD002971.pub6. PMID 39239939
- [Background] Quigley M, Embleton ND, McGuire W. Formula versus donor breast milk for feeding preterm or low birth weight infants. Cochrane Database Syst Rev. 2019 Jul 19;7(7):CD002971. doi: 10.1002/14651858.CD002971.pub5. PMID 31322731
- [Background] Quigley M, McGuire W. Formula versus donor breast milk for feeding preterm or low birth weight infants. Cochrane Database Syst Rev. 2014 Apr 22;(4):CD002971. doi: 10.1002/14651858.CD002971.pub3. PMID 24752468
- [Background] Hair AB, Peluso AM, Hawthorne KM, Perez J, Smith DP, Khan JY, O'Donnell A, Powers RJ, Lee ML, Abrams SA. Beyond Necrotizing Enterocolitis Prevention: Improving Outcomes with an Exclusive Human Milk-Based Diet. Breastfeed Med. 2016 Mar;11(2):70-4. doi: 10.1089/bfm.2015.0134. Epub 2016 Jan 20. PMID 26789484
- [Background] Walsh MC, Kliegman RM. Necrotizing enterocolitis: treatment based on staging criteria. Pediatr Clin North Am. 1986 Feb;33(1):179-201. doi: 10.1016/s0031-3955(16)34975-6. PMID 3081865
- [Background] Bell MJ, Ternberg JL, Feigin RD, Keating JP, Marshall R, Barton L, Brotherton T. Neonatal necrotizing enterocolitis. Therapeutic decisions based upon clinical staging. Ann Surg. 1978 Jan;187(1):1-7. doi: 10.1097/00000658-197801000-00001. PMID 413500
- [Background] Ruiz-Giardin JM, Ochoa Chamorro I, Velazquez Rios L, Jaqueti Aroca J, Garcia Arata MI, SanMartin Lopez JV, Guerrero Santillan M. Blood stream infections associated with central and peripheral venous catheters. BMC Infect Dis. 2019 Oct 15;19(1):841. doi: 10.1186/s12879-019-4505-2. PMID 31615450
- [Background] Heilmann C, Ziebuhr W, Becker K. Are coagulase-negative staphylococci virulent? Clin Microbiol Infect. 2019 Sep;25(9):1071-1080. doi: 10.1016/j.cmi.2018.11.012. Epub 2018 Nov 29. PMID 30502487
- [Background] Shalabi M, Adel M, Yoon E, Aziz K, Lee S, Shah PS; Canadian Neonatal Network. Risk of Infection Using Peripherally Inserted Central and Umbilical Catheters in Preterm Neonates. Pediatrics. 2015 Dec;136(6):1073-9. doi: 10.1542/peds.2015-2710. Epub 2015 Nov 16. PMID 26574592
- [Background] Marchant EA, Boyce GK, Sadarangani M, Lavoie PM. Neonatal sepsis due to coagulase-negative staphylococci. Clin Dev Immunol. 2013;2013:586076. doi: 10.1155/2013/586076. Epub 2013 May 22. PMID 23762094
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Background] Janes M, Kalyn A, Pinelli J, Paes B. A randomized trial comparing peripherally inserted central venous catheters and peripheral intravenous catheters in infants with very low birth weight. J Pediatr Surg. 2000 Jul;35(7):1040-4. doi: 10.1053/jpsu.2000.7767. PMID 10917292
- [Background] Bjorkman L, Ohlin A. Scrubbing the hub of intravenous catheters with an alcohol wipe for 15 sec reduced neonatal sepsis. Acta Paediatr. 2015 Mar;104(3):232-6. doi: 10.1111/apa.12866. Epub 2015 Jan 30. PMID 25399485
- [Background] Payne V, Hall M, Prieto J, Johnson M. Care bundles to reduce central line-associated bloodstream infections in the neonatal unit: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F422-F429. doi: 10.1136/archdischild-2017-313362. Epub 2017 Nov 25. PMID 29175985
- [Background] Flannery DD, Edwards EM, Coggins SA, Horbar JD, Puopolo KM. Late-Onset Sepsis Among Very Preterm Infants. Pediatrics. 2022 Dec 1;150(6):e2022058813. doi: 10.1542/peds.2022-058813. PMID 36366916
- [Background] Miller J, Tonkin E, Damarell RA, McPhee AJ, Suganuma M, Suganuma H, Middleton PF, Makrides M, Collins CT. A Systematic Review and Meta-Analysis of Human Milk Feeding and Morbidity in Very Low Birth Weight Infants. Nutrients. 2018 May 31;10(6):707. doi: 10.3390/nu10060707. PMID 29857555
- [Background] Arslanoglu S, Boquien CY, King C, Lamireau D, Tonetto P, Barnett D, Bertino E, Gaya A, Gebauer C, Grovslien A, Moro GE, Weaver G, Wesolowska AM, Picaud JC. Fortification of Human Milk for Preterm Infants: Update and Recommendations of the European Milk Bank Association (EMBA) Working Group on Human Milk Fortification. Front Pediatr. 2019 Mar 22;7:76. doi: 10.3389/fped.2019.00076. eCollection 2019. PMID 30968003
- [Background] Gregory KE, Samuel BS, Houghteling P, Shan G, Ausubel FM, Sadreyev RI, Walker WA. Influence of maternal breast milk ingestion on acquisition of the intestinal microbiome in preterm infants. Microbiome. 2016 Dec 30;4(1):68. doi: 10.1186/s40168-016-0214-x. PMID 28034306
- [Background] Cong X, Judge M, Xu W, Diallo A, Janton S, Brownell EA, Maas K, Graf J. Influence of Feeding Type on Gut Microbiome Development in Hospitalized Preterm Infants. Nurs Res. 2017 Mar/Apr;66(2):123-133. doi: 10.1097/NNR.0000000000000208. PMID 28252573
- [Background] Levy I, Comarsca J, Davidovits M, Klinger G, Sirota L, Linder N. Urinary tract infection in preterm infants: the protective role of breastfeeding. Pediatr Nephrol. 2009 Mar;24(3):527-31. doi: 10.1007/s00467-008-1007-7. Epub 2008 Oct 21. PMID 18936982
- [Background] Mohseny AB, van Velze V, Steggerda SJ, Smits-Wintjens VEHJ, Bekker V, Lopriore E. Late-onset sepsis due to urinary tract infection in very preterm neonates is not uncommon. Eur J Pediatr. 2018 Jan;177(1):33-38. doi: 10.1007/s00431-017-3030-9. Epub 2017 Oct 23. PMID 29063210
- [Background] Downey LC, Benjamin DK Jr, Clark RH, Watt KM, Hornik CP, Laughon MM, Cohen-Wolkowiez M, Smith PB. Urinary tract infection concordance with positive blood and cerebrospinal fluid cultures in the neonatal intensive care unit. J Perinatol. 2013 Apr;33(4):302-6. doi: 10.1038/jp.2012.111. Epub 2012 Aug 30. PMID 22935772
- [Background] Carl MA, Ndao IM, Springman AC, Manning SD, Johnson JR, Johnston BD, Burnham CA, Weinstock ES, Weinstock GM, Wylie TN, Mitreva M, Abubucker S, Zhou Y, Stevens HJ, Hall-Moore C, Julian S, Shaikh N, Warner BB, Tarr PI. Sepsis from the gut: the enteric habitat of bacteria that cause late-onset neonatal bloodstream infections. Clin Infect Dis. 2014 May;58(9):1211-8. doi: 10.1093/cid/ciu084. Epub 2014 Mar 18. PMID 24647013
- [Background] Goldblum RM, Schanler RJ, Garza C, Goldman AS. Human milk feeding enhances the urinary excretion of immunologic factors in low birth weight infants. Pediatr Res. 1989 Feb;25(2):184-8. doi: 10.1203/00006450-198902000-00021. PMID 2919134
- [Background] Nangia S, Vadivel V, Thukral A, Saili A. Early Total Enteral Feeding versus Conventional Enteral Feeding in Stable Very-Low-Birth-Weight Infants: A Randomised Controlled Trial. Neonatology. 2019;115(3):256-262. doi: 10.1159/000496015. Epub 2019 Jan 30. PMID 30699425